CLINICAL TRIAL: NCT03977181
Title: Leveraging Community-based Platforms to Improve Access and Adherence to PrEP for Young Women in South Africa
Brief Title: The Community PrEP Study to Assess the Acceptance of PrEP Delivered Through CBCT Platforms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Professional Development (Pty) Ltd (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH); Desmond Tutu HIV Centre (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH114648 (NIH); 1R01MH114648 (NIH)
Record Dates: First submitted 2019-05-23; First posted 2019-06-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: PrEP; HIV Prevention; Adolescence; Cost-effectiveness
Keywords: PrEP; HIV Prevention; Adherence Support; Adolescence; South Africa

STUDY DESIGN:
Intervention Model Description: Investigators will perform a 3-arm randomized controlled trial, with participants randomized to one of the following arms: Arm 1) a group-based community health club akin to an ART adherence club; Arm 2) one-on-one adherence counseling and support; or Arm 3) community-based medication dispensary.
Masking Description: The allocation of study arm is concealed to study staff during randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Club (Experimental): A group-based community health club akin to an ART adherence club
  Interventions: Behavioral: Group-based Community Health Club
- One-on-one (Experimental): One-on-one adherence counselling and support
  Interventions: Behavioral: Individual-based Adherence Support
- Medication pick-up (No Intervention): Community-based medication dispensary

INTERVENTIONS:
Behavioral: Group-based Community Health Club — GBHCs will be facilitated by trained Lay Health Counsellors (LHC). GBHCs will consist of a maximum 20 participants. GBHC sessions will held multiple times a month in each study area, allowing for flexibility for study participants. Sessions will be held at a safe and secure, centrally located area within the study community, and will be regularly monitored and assessed by the study coordinator. Participants will be invited to join a club-specific WhatsApp group to facilitate group communication and adherence support throughout the month. They will also be invited to partner up with another participant to provide mutual peer support. Permission will be sought from group-based adherence support participants before they are added to WhatsApp groups. Group adherence counsellors assigned will be members of WhatsApp groups, and will monitor all shared content to ensure that no inappropriate content or private information is shared in the group.
  Arms: Health Club
Behavioral: Individual-based Adherence Support — IAS participants will be matched to a LHC and will schedule IAS sessions once-a-month for the duration of the study. These sessions will be held at a centralized location within the study community. The sessions will be semi-structured to allow for participant-driven discussion of any adherence challenges and key-messages. The adherence curriculum will also explore motivations for PrEP and adherence and focus on practical adherence tips, environmental cues, integration of PrEP within daily routines, short-term goal-setting, problem-solving, safe PrEP disclosure and social support, risk reduction counselling, partner communication, and HIV risk perception. A subset of IAS sessions will be audio-recorded for quality assurance by investigators and the study coordinator. These recordings are for training purposes only and will not form part of the dataset. Consent for recording IAS sessions will be sought from participants during the pre-enrolment consent process.
  Arms: One-on-one

SUMMARY:
The investigators aim to 1) speed up access to and delivery of PrEP to young women, and 2) compare interventions to support and maximize the prevention-effective use of PrEP. Specifically, the investigators aim to answer the following two questions: 1) how can the study use existing community-based platforms to identify and deliver PrEP to those in need? and 2) which adherence support interventions are most likely to engender effective use of PrEP? The investigators propose to answer these questions by leveraging existing community-based HIV testing platforms in South Africa and use a mixed methods approach to optimize the PrEP cascade and evaluate a community-based PrEP adherence program for young women.

DETAILED DESCRIPTION:
Worldwide, about 1.9 million people became infected with HIV in 2015, most of whom live in Southern and East Africa. In South Africa, the HIV incidence rate among young women ages 15-24 (2.5%) is four times higher than their male counterparts (0.6%). Recent HIV prevention trials in South Africa documented incidence rates of 5-6% per year in 15-24 year old young women. Given this high incidence of HIV, implementing effective HIV prevention strategies - including PrEP - is crucial to controlling HIV globally.

The proposed study leverages existing community-based HIV counseling and testing platforms in South Africa and evaluates, using a mixed methods approach, a community-based PrEP adherence program for young women whilst optimizing the PrEP cascade. Numerous barriers have been described that delay or block young women from accessing clinic-based health services, especially reproductive health and HIV testing and prevention services. Consequently, reaching young women at large scale with HIV prevention services requires delivery platforms outside of clinic-based facilities. Community-based counseling and testing programs have shown the greatest coverage and potential to achieve high levels of knowledge of HIV serostatus and linkage to HIV care. Using community-based counseling and testing programs, this proposal will deliver PrEP as part of a population-level combination prevention program, which is necessary to substantially reduce HIV incidence.

The investigators propose to answer key research questions through the following; Specific Aims: 1) Assess young women's uptake of PrEP when delivered through large-scale community-based HIV counseling and testing platforms in urban and rural settings in South Africa, 2) Evaluate community-based scalable interventions to achieve prevention-effective adherence to PrEP among young women, and 3) Evaluate the cost per young woman initiated on PrEP and provided adherence support through community-based platforms, and the cost-effectiveness per incident HIV infection averted. In order to achieve Aim 1, the study will leverage from on-going, at-scale CBCT programs and platforms (mobile unit and systematic home-based testing) to identify and link young women to community-based PrEP initiation services. In order to achieve Aim 2, the study will perform a 3-arm randomized controlled trial, with participants randomized to one of the following arms: Arm 1) a group-based community health club akin to an ART adherence club; Arm 2) one-on-one adherence counseling and support; Arm 3) community-based medication dispensary.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as female (regardless of assigned sex at birth)
* 16 - 25 years of age.
* HIV negative (confirmed during CBCT testing)
* At risk for HIV acquisition
* Express interest in taking PrEP

Exclusion Criteria:

* Planning to relocate in the next 12 months
* Positive HIV test at screening or enrolment
* Pregnant
* Breastfeeding
* Current participation in other HIV prevention studies (clinical or behavioural)
* Current use of ARV drugs for post-exposure prophylaxis (PEP)
* Presence of any disease or health condition, self-reported or identified by initiation clinician, that may prevent participation.

Ages: 16 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identified as female (regardless of assigned sex at birth)
Enrollment: 480 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
The cost per adolescent girl and young women on pre-exposure prophylaxis | 10 months
  Itemized cost menus
The incremental cost-effectiveness ratio per incidence HIV case averted | 10 months
  Dynamic infectious disease model of HIV

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Medina-Marino, PhD, Principal Investigator — Foundation for Professional Development; Linda-Gail Bekker, MBChB, DTMH, DCH, FCP, PhD, Principal Investigator — Desmund Tutu HIV Centre
Locations (1):
- Buffalo City Metro, East London, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, Analytic Code
Access Criteria: Based on contractual agreement

REFERENCES:
- [Derived] de Vos L, Krogstad Mudzingwa E, Fynn L, Atujuna M, Webb Mazinyo E, Kodi K, Hosek S, Katz IT, Celum C, Bekker LG, Daniels J, Medina-Marino A. Study-to-Clinic Transition and Daily Oral PrEP Access Experiences Among AGYW in Eastern Cape, South Africa: Insights from the Community PrEP Study. AIDS Behav. 2025 Aug;29(8):2574-2587. doi: 10.1007/s10461-025-04718-7. Epub 2025 Apr 17. PMID 40240718
- [Derived] Krogstad Mudzingwa E, de Vos L, Atujuna M, Fynn L, Mugore M, Mabandla S, Hosek S, Celum C, Bekker LG, Daniels J, Medina-Marino A. High study participation but diverging adherence levels: qualitatively unpacking PrEP use among adolescent girls and young women over two years in Eastern Cape, South Africa. J Behav Med. 2024 Apr;47(2):320-333. doi: 10.1007/s10865-023-00462-2. Epub 2023 Dec 11. PMID 38081955
- [Derived] de Vos L, Mudzingwa EK, Fynn L, Atujuna M, Mugore M, Gandhi M, Celum C, Hosek S, Bekker LG, Daniels J, Medina-Marino A. Factors that influence adolescent girls and young women's re-initiation or complete discontinuation from daily oral PrEP use: a qualitative study from Eastern Cape Province, South Africa. J Int AIDS Soc. 2023 Sep;26(9):e26175. doi: 10.1002/jia2.26175. PMID 37758649
- [Derived] Mudzingwa EK, de Vos L, Atujuna M, Fynn L, Mugore M, Hosek S, Celum C, Bekker LG, Daniels J, Medina-Marino A. Factors influencing adolescent girls and young women's uptake of community-based PrEP services following home-based HIV testing in Eastern Cape, South Africa: a qualitative study. AIDS Behav. 2022 Nov;26(11):3726-3739. doi: 10.1007/s10461-022-03702-9. Epub 2022 Jun 2. PMID 35653046
- [Derived] Medina-Marino A, Bezuidenhout D, Hosek S, Barnabas RV, Atujuna M, Bezuidenhout C, Ngwepe P, Peters RPH, Little F, Celum CL, Daniels J, Bekker LG. The Community PrEP Study: a randomized control trial leveraging community-based platforms to improve access and adherence to pre-exposure prophylaxis to prevent HIV among adolescent girls and young women in South Africa-study protocol. Trials. 2021 Jul 26;22(1):489. doi: 10.1186/s13063-021-05402-6. PMID 34311754